CLINICAL TRIAL: NCT02283970
Title: Investigation of Patients With BAV Requiring Valve and/or Aortic Repair. Correlation of Surgical and ECO Distinctive Features With Histologic and Genetic Findings in Phenotypically Homogeneous Outlier Cases (GISSI VAR)
Brief Title: Investigation of Patients With BAV Requiring Valve and/or Aortic Repair (GISSI Outliers VAR)
Acronym: VAR
Status: Completed | Type: Observational
Sponsor: Gruppo di Ricerca GISSI (Other)
Responsible Party: Sponsor
Other Study IDs: K11
Record Dates: First submitted 2014-10-17; First posted 2014-11-05 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Bicuspid Aortic Valve; Aortic Regurgitation; Aortic Dilatation
MeSH Terms: conditions — Bicuspid Aortic Valve Disease; Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples and tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- BAV and aortic regurgitation: BAV Diagnosis, Aortic Regurgitation with surgical indication (according to current clinical guidelines or best clinical practice), normal ascending aorta
- BAV and Ascending aorta dilatation: BAV diagnosis, no or trivial Aortic Regurgitation, ascending aorta dilatation with surgical indication (according to current clinical guidelines or best clinical practice)
- BAV, aortic regurgitation and dilatation: BAV diagnosis, Aortic Regurgitation and ascending aorta dilatation with surgical indication (according to current clinical guidelines or best clinical practice).
- BAV with aortic stenosis in pts>60yrs: BAV diagnosis, Aortic stenosis with surgical indication (according to current clinical guidelines or best clinical practice). Normal ascending aorta

SUMMARY:
Prospective longitudinal study on four small groups of surgical patients affected by: BAV with isolated regurgitation, BAV associated with aorta dilatation, or both and BAV with isolated stenosis in over 60 year-old patients.

The aim of the study is to select homogeneous small groups of surgical patients with the same subtype of BAV and same aortic behaviour and identify markers/predictors of favorable-unfavorable aortic wall evolution to evaluate if there is a BAV phenotype more likely to be considered at high risk for aortic degeneration.

DETAILED DESCRIPTION:
The aim of the study is to select homogeneous small groups of surgical patients with the same subtype of BAV and same aortic behaviour and identify markers/predictors of favorable-unfavorable aortic wall evolution to evaluate if there is a BAV phenotype more likely to be considered at high risk for aortic degeneration. The study will focus on multiple aspects of BAV disease. What follows will be considered and combined:

Aortic valve, aorta root and ascending aorta morphology The use of two- (2DE) and three-dimensional (3DE) trans-thoracic (TTE) and/or transoesophageal (TOE) echocardiography can identify all kind of BAV morphology (leaflet position and coronary ostia displacement). It also gives quali- quantitative information about root and ascending aorta morphology and size.

BAV genetics Recently, missense mutations in the NOTCH1 gene have been shown to be associated with calcific aortic valve disease plus BAV. However mutations in the NOTCH1 gene only partially explain the presence of BAV in the absence of other syndromic diseases (i.e. Marfan Syndrome, Loeys Dietz Syndrome type I and II and Ehlers Danlos type IV Syndrome).

BAV Histology In all enrolled patients, during operation, tissue samples will be collected from valve cusps (in case of valve involvement), aortic wall (aortic root, concavity or convexity of ascending aorta) or from both of them. Samples will be analyzed in order to classify medial and intimal disruption and changes.

Study Design and Setting of the Study The first step will consist in enrolling patients with echocardiographic diagnosis of BAV and indication for surgery. From the echo data, aortic valve, as well as aortic root and ascending aorta morphology will be assessed in order to classify patients in each phenotypic pattern. The echo images from participating centres will be sent to an echo core lab for quali- quantitative analysis (see below) and all data will be recorded in a specific database.

The second step will consider first-degree relatives of each enrolled patient. The investigators will ask every first degree relative to perform a screening TTE in order to find out, according to familiar aetiology of BAV, the presence of BAV and/or associated disease (aortic root or ascending aorta enlargement or coronary ostia displacement).

The third step will consist in collecting blood samples from each patient and from any of first-degree relatives with BAV diagnosis. BAV-specific genetic tests will be performed and all data will be recorder in a specific database.

The fourth intraoperative step will consist in :

1. performing a 3D TOE in order to study the geometry and the dynamic behaviour of the aortic valve and root and
2. in collecting surgical tissue samples: during operation there will be described precisely the anatomy of the valve and the aorta in detail; then, from the usual site of surgery, there will be collected valve and aortic wall samples in order to perform histological, immunohistochemical and genetics tests.

Blood and surgical samples will be stored in a bio-bank for future analysis related to this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years-old and under the age of 60 (age selection will prevent from enrolling patient with age-related valve and aortic wall degeneration). For the BAV stenosis group there will be considered patients over 60 years-old: including the most frequent form of BAV disease and the commonest age, this group could be used as a control group compared to the outlier ones.
* Echo diagnosis of BAV and indication to surgery:

BAV with isolated regurgitation, BAV with normal valvular function but associated aorta dilatation, BAV with both valve regurgitation and aortic dilatation BAV with isolated stenosis

- Signed informed consent

Exclusion Criteria:

* Patient with a previous cardiac or great vessels surgery
* coexistent coarctation of the aorta
* non-associated cardiac diseases: valve disease (other than aortic), ischemic disease, congenital heart disease.
* Marfan syndrome or other connective tissue disorders involving aortic valve and aortic wall disease (history of disease or clinical signs).
* Other conditions/circumstances likely to lead to poor study adherence (e.g. psychological or organizational reasons).
* Serious disease other than aortic, severely limiting life expectancy.
* Patients who refuse to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: BAV patients eligible for cardiac surgery due to each of these conditions: BAV Regurgitation isolated, ascending aorta aneurysm in normal BAV or both AR and ascending aorta aneurysm, BAV stenosis isolated in over 60 year-old patients.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2012-12; Primary Completion 2014-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Mutation in NOTCH1 gene | Enrollment
  The strongest causative gene associated with BAV is NOTCH1. Its 34 coding exons will be sequenced to search for variants likely to be causative.
  The presence of sequence variation will be confirmed using a different method, starting from a new amplification (RFLP or High Resolution Melting-HRM). The pathogeneticity of the mutation will be evaluated screening 500 DNA controls (1000 chromosomes) to estimate the alleles' frequencies (HRM; ABI Prism 7900HT). Finally a familial segregation analysis will be performed to verify the association with the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Attilio Maseri, MD, Study Chair — Dondazione per il Tuo cuore-HCF Onlus
Locations (10):
- Italy (10):
  - Casa Di Cura Villa Sant'Anna, Catanzaro, CZ
  - Aou Careggi, Florence, FI
  - Ospedale San Raffaele, Milan, MI
  - Centro Cardiologico Monzino, Milan, MI
  - Ospedale Niguarda, Milan, MI
  - Irccs Policlinico San Donato, San Donato Milanese, MI
  - Aou Santa Maria Della Misericordia, Udine, UD
  - Ospedale Dell'Angelo, Mestre, VE
  - Ospedale San Camillo, Roma
  - Azienda Osp. Univ. S. Giovanni Battista, Torino

REFERENCES:
- [Background] Merlanti B, De Chiara B, Maggioni AP, Moreo A, Pileggi S, Romeo G, Russo CF, Rizzo S, Martinelli L, Maseri A; VAR Study Group. Rationale and design of GISSI OUTLIERS VAR Study in bicuspid aortic valve patients: prospective longitudinal, multicenter study to investigate correlation between surgical, echo distinctive features, histologic and genetic findings in phenotypically homogeneous outlier cases. Int J Cardiol. 2015 Nov 15;199:180-5. doi: 10.1016/j.ijcard.2015.06.182. Epub 2015 Jul 6. PMID 26197404